CLINICAL TRIAL: NCT04018625
Title: An Internet-Delivered Mind-Body Program for Reducing Prenatal Maternal Stress
Brief Title: The Stony Brook University Calm-Mom Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Massachusetts General Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Brittain Lynn Mahaffey, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 972565-4; K23HD092888 (NIH)
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pregnancy Related; Stress, Psychological; Anxiety; Perinatal Depression
Keywords: Prenatal Maternal Stress; Perinatal Mental Health; Pregnancy; Perinatal Anxiety; Perinatal Depression
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Intervention versus treatment as usual.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants (n = 30) will be randomized to receive the SMART Pregnancy stress management program via an online portal.
  Interventions: Behavioral: SMART Mom
- Treatment as usual (Active Comparator): Participants (n = 30) will be randomized to receive treatment as usual, including referrals to community based support groups and individual mental health providers.
  Interventions: Behavioral: Mama Support

INTERVENTIONS:
Behavioral: SMART Mom — SMART Pregnancy is an 8-session online stress management program offered in a group format. SMART Pregnancy is an adaptation of the Stress Management and Resiliency Training Program (Park et al., 2012).
  Arms: Intervention
Behavioral: Mama Support — Participants will be enrolled in an 8-week time and attention matched, process-based support group.
  Arms: Treatment as usual

SUMMARY:
The present trial will evaluate the feasibility, acceptability and preliminary efficacy of 2 different internet-delivered programs for prenatal maternal stress. The Stress Managment and Resiliency Training Program (SMART-Mom program), an 8-session Cognitive Behavior Therapy (CBT) based mind body program and the Mama Support Program, an 8-session social support group program. Sixty pregnant women (<20 weeks Estimated Gestational Age) will be screened and either enrolled in the online SMART Mom Program or the Mama Support Program. Outcomes, including maternal perceived stress, depression, and anxiety will be assessed at post-treatment, three, and six months post program completion. Potential impact on infant health outcomes will be assessed via post-delivery electronic medical record review.

DETAILED DESCRIPTION:
Aim 1: The investigators will conduct a randomized clinical trial (RCT; n=60) to assess the feasibility, acceptability and preliminary efficacy of the Stress Management and Resillency Training program (SMART Pregnancy) delivered online versus a time and attention matched prenatal support group (Mama Support). It is expected that SMART-pregnancy participants will demonstrate high levels of treatment engagement and adherence. It is predicted that participants in the SMART-Pregnancy condition will demonstrate improvements in emotional distress and stress regulation (as indexed by hair cortisol concentrations) at post-treatment and 3 month follow-up. Aim 2: The investigators will conduct a postnatal chart review to explore secondary treatment benefits including pre-and postnatal maternal health and birth outcomes.

ELIGIBILITY:
Inclusion Criteria:

* <21 weeks pregnant with medically confirmed viability
* Speak, read and write in English fluently,
* Endorse elevated levels of prenatal maternal stress (PNMS; i.e., New Prenatal Distress Questionnaire Score > 19).

Exclusion Criteria:

* Current enrollment in individual or group psychotherapy
* Current un-managed serious mental illness including bipolar disorder and psychosis
* History of previous suicide attempt
* Inappropriate for participation in group therapy format as determined by study director

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress as indexed by Perceived Stress Scale (PSS) score | baseline, 8 weeks post enrollment, 20 weeks post enrollment
  Gold standard measure of subjective stress experiences. Total scores range from 0 to 40; higher scores indicate greater stress.
Change in prenatal maternal distress as indexed by Prenatal Distress Questionnaire (NuPDQ) score | baseline, 8 weeks post enrollment
  Measure of prenatal maternal distress. Total scores range form 0-35; higher scores indicate greater pregnancy-related distress.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) V.1 Emotional Distress-Depression | baseline, 8 weeks post enrollment, 20 weeks post enrollment
  Standardized depression symptom measure. Total scores range from 8-40; higher values represent greater distress/depression.
Patient-Reported Outcomes Measurement Information System (PROMIS) V.1 Emotional Distress-Anxiety | baseline, 8 weeks post enrollment, 20 weeks post enrollment
  Standardized anxiety symptom measure. Total scores range from 6-30; higher values represent greater anxiety.
Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | baseline, 8 weeks post enrollment, 20 weeks post enrollment
  Widely used mindfulness measure; total scores range from 12-60; higher scores represent greater mindfulness.
Measure of Current Status-Form A (MOCS-A) | baseline, 8 weeks post enrollment, 20 weeks post enrollment
  Measure of stress-related coping. Total scores range from 0-52; higher scores represent better coping.

OTHER OUTCOMES:
Birthweight | Chart review occurring at 6 week postpartum visit.
  Infant weight (in grams) at birth.
Gestational Age | Chart review occurring at 6 week postpartum visit.
  Infant gestational age (in weeks) at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Brittain L Mahaffey, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Department of Psychiatry, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators are committed to sharing the research data that is generated in this proposal. Research data will be shared according to NIH guidelines. All research data is collected and stored in accordance with HIPAA compliance, and any shared datasets resulting from human participant research will be free of any identifiers that would allow disclosure of individual subjects.
Supporting Information: Study Protocol, SAP
Time Frame: Timelines for distribution of data will vary, however the study team will make every effort to make data available in a timely fashion. It is expected that data from this proposal will presented at scientific meetings, and publications will be made available through PubMed Central no later than 12 months after publication.
Access Criteria: The data will be available to users under a data sharing agreement that includes a commitment to: 1) using the data for research purposes only, 2) properly securing the data in accordance with HIPAA compliance requirements, and 3) destroying the data after analyses are completed.
URL: http://publicaccess.nih.gov/policy.htm